CLINICAL TRIAL: NCT02501382
Title: Biomarkers in Necrotizing Soft Tissue Infections - Effects of Hyperbaric Oxygen Treatment on the Immune Response
Brief Title: Modulation of Biomarkers in Patients With Flesh-eating Bacterial Infections After With Hyperbaric Oxygen Treatment
Acronym: BIONEC-II
Status: Completed | Type: Observational
Sponsor: Ole Hyldegaard (Other)
Responsible Party: Sponsor-Investigator, Ole Hyldegaard, MD, PhD, DMSci, Rigshospitalet, Denmark
Organization: Rigshospitalet, Denmark (Other)
Other Study IDs: BIONEC2-MBH-2015
Record Dates: First submitted 2015-07-03; First posted 2015-07-17 (Estimated); Last update posted 2019-06-24 (Actual); Status verified 2019-06

CONDITIONS: Necrotizing Soft Tissue Infection; Necrotizing Fasciitis; Gas Gangrene; Fournier Gangrene
Keywords: Fasciitis; Fasciitis, Necrotizing; Soft tissue infections; Fournier's gangrene; Immunopathogenesis
MeSH Terms: conditions — Fasciitis, Necrotizing; Gas Gangrene; Fournier Gangrene; Fasciitis; Soft Tissue Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Whole blood and plasma/serum
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Patients with NSTI treated with HBOT: NSTI definition: An infection that requires acute hospitalization with intensive care treatment and/or surgery as a consequence of severe soft tissue infection causing necrosis in subcutis, muscle and/or fascia.

SUMMARY:
The purpose of this study is to investigate the effects of hyperic oxygen treatment on the immune response in patients with necrotizing soft tissue infections

DETAILED DESCRIPTION:
Necrotizing soft tissue infections (NSTI) is a complex, multi-factorial disease and the bacteria show a diverse microbial etiology. The exentisive inflammatory response caused by these bacteria is thought to be a main course of death. In Denmark, most NSTI patients are treated with hyperic oxygen therapy (HBOT). However, the effects of HBOT have never been investigated in NSTI patients.

Location: Copenhagen University Hospital, Rigshospitalet, Denmark.

Design: Observational cohort study.

Cohort: NSTI patients in Denmark treated with HBOT.

Biomarkers: Cytokines, acute-phase proteins, vasoactive biomarkers and other inflammatory biomarkers.

Sample size calculation: The investigators expect a mean IL-6 concentration before HBOT of 3500 pg/ml (standard deviation 1500 pg/ml) and consider a reduction of 800 pg/ml to be clinically relevant. With an alpha = 0.05 and a power of 80%, 112 patients will be required.

Data: The Danish Data Protection Agency has approved the processing of personal data for the NSTI patients (J. no. 30-0900).

Ethics: The trial will adhere to the Helsinki Declaration and the Danish law. The National Ethics Committee and the Regional Scientific Ethics Committee of Copenhagen have approved the study (CVK-1211709 and H-2-2014-071).

Analysis: Biomarker analyses will be performed once the recruitment of patients has ended.

ELIGIBILITY:
Inclusion criteria:

* Necrotizing soft tissue infection based on surgical findings
* Admitted to/planned to be admitted to the ICU at Rigshospitalet and/or operated for NSTI at Rigshospitalet
* Receving a minimum of 1 HBOT

Exclusion criteria:

* Patients who at the operating theatre were categorized as a non-NSTI patient

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with NSTI treated with HBOT
Sampling Method: Probability Sample
Enrollment: 65 (Actual)
Dates: Start 2013-02 (Actual); Primary Completion 2015-12-01 (Actual); Study Completion 2015-12-01 (Actual)

PRIMARY OUTCOMES:
IL-6 as a marker of treatment effects after HBOT | Change from baseline in IL-6 concentration after first HBOT administered during the first 24 hours of admission

SECONDARY OUTCOMES:
Inflammatory biomarkers as indicators of treatment effects after HBOT | The first 5 days of admission
Vasoactive biomarkers as indicators of treatment effects after HBOT | The first 5 days of admission
Mortality | 30, 90, 180 days
Amputation rate | During the first 7 days of ICU admission
SAPS II assessment | During the first 24 hours of ICU admission
APACHE II assessment | During the first 7 days of ICU admission
SOFA score assessment | During the first 7 days of ICU admission
Anaya score assessment | During the first 7 days of ICU admission
LRINEC score assessment | During the first 7 days of ICU admission
Multiple organ failure assessed by the MODS score | During the first 7 days of ICU admission
Number of debridements | During the first 7 days of ICU admission
Microbial etiology results from blood and tissue samples | During the first 7 days of ICU admission

CONTACTS AND LOCATIONS:
Overall Officials: Ole Hyldegaard, MD, PhD, Study Director — Department of Anaesthesiology, Center of Hyperbaric Treatment, sect. 4092, Copenhagen University Hospital, Denmark; Marco Bo Hansen, MD, Principal Investigator — Department of Anaesthesiology, Center of Hyperbaric Treatment, sect. 4092, Copenhagen University Hospital, Denmark
Locations (1):
- Copenhagen University Hospital, Rigshospitalet, Copenhagen, Denmark